CLINICAL TRIAL: NCT02161614
Title: Flow-mediated Evaluation of the Brachial Artery of Climacteric Women Using Estradiol Valerate and Placebo. Randomized, Double Blinded, Placebo Controlled Study.
Brief Title: Vascular Effect of Estradiol Valerate Versus Placebo Evaluated by Flow-mediated Dilatation of Brachial Artery
Acronym: VEDILA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Selmo Geber, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DILA V E2
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Flow-mediated Dilation Evaluation of the Brachial Artery
Keywords: hormone replacement therapy; Dopplervelocimetry; Flow-mediated dilation; menopause; Estradiol valerate
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will use placebo for 30 days
  Interventions: Drug: Placebo
- Estradiol Valerate (Experimental): patients will use estradiol valerate 1mg/day during 30 days
  Interventions: Drug: Estradiol valerate

INTERVENTIONS:
Drug: Estradiol valerate
  Arms: Estradiol Valerate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the vascular effects of estradiol valerate on climacteric women measured by flow-mediated evaluation of the brachial artery using high resolution ultrasound and compare to placebo.

DETAILED DESCRIPTION:
The interruption of the secretion of sex steroids that occurs after menopause, determines a change in vascular pattern at various levels. As a result, several side effects might appear and interfere with women's quality of life and health. The use of hormone replacement therapy has contributed to the improvement in these effects. It has been observed vascular beneficial effects of sex steroids in premenopausal women, and of hormone replacement therapy (HRT) in climacteric women, on the central retinal arteries. The objective of this study is to evaluate the effects of estradiol valerate on flow-mediated dilation of the brachial artery.

ELIGIBILITY:
Inclusion Criteria:

* Women without menstrual cycles within the last 12 months and follicle stimulating hormone (FSH)>30International Units / Liter
* Healthy women
* Women that were not using drugs with potential vascular effect within the last 1 year
* Women that never used hormone replacement therapy

Exclusion Criteria:

* Smoking
* Blood Pressure > 160/90 mm Hg.
* Breast and or endometrial cancer
* History of acute myocardial infarction
* Diabetes
* Vaginal bleeding of any origin
* Hepatic disease
* thrombophlebitis or thromboembolic disorders

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the brachial artery | 30 days after treatment started

CONTACTS AND LOCATIONS:
Overall Officials: Selmo Geber, MD PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Hospital das Clinicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Faria AF, de Souza MA, Geber S. Vascular resistance of central retinal artery is reduced in postmenopausal women after use of estrogen. Menopause. 2011 Aug;18(8):869-72. doi: 10.1097/gme.0b013e31820cc60c. PMID 21471823